CLINICAL TRIAL: NCT02580669
Title: Study by Magnetic Resonance Imaging of the Modifications of the Vasoreactivity and Cerebral Connectivity in the Progressive Forms of Multiple Sclerosis
Brief Title: Study by Magnetic Resonance Imaging in the Progressive Forms of Multiple Sclerosis
Acronym: VASOSEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion period ended
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 9090
Record Dates: First submitted 2015-09-25; First posted 2015-10-20 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Progressive Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis, Relapsing-Remitting | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Progressive Multiple Sclerosis (Experimental): 22 patients with Progressive Multiple Sclerosis will be included and they get an Neuropsychological assessment, a Neurologic consultation and MRIs (with vasoreactivity testing)
  Interventions: Other: Neuropsychological assessment; Other: Neurologic consultation; Other: MRIs (with vasoreactivity testing)
- Multiple Sclerosis, Relapsing-Remitting (Experimental): 22 patients with Multiple Sclerosis, Relapsing-Remitting will be included and they get an Neuropsychological assessment, a Neurologic consultation and MRIs (with vasoreactivity testing)
  Interventions: Other: Neuropsychological assessment; Other: Neurologic consultation; Other: MRIs (with vasoreactivity testing)
- Healthy volunteers (22 patients) (Experimental): 22 healthy volunteers will be included and they get an Neuropsychological assessment and MRIs (with vasoreactivity testing)
  Interventions: Other: Neuropsychological assessment; Other: MRIs (with vasoreactivity testing)

INTERVENTIONS:
Other: Neuropsychological assessment — A neuropsychological assessment is done
Other: Neurologic consultation — A neurologic consultation is done
  Arms: Multiple Sclerosis, Relapsing-Remitting; Progressive Multiple Sclerosis
Other: MRIs (with vasoreactivity testing) — MRIs (with vasoreactivity testing) is done

SUMMARY:
The goal of this study is to show pattern differences of vasoreactivity and connectivity between Progressive Multiple Sclerosis and Relapsing Remitting Multiple Sclerosis, by the use of methods of advanced brain MRIs and the Diffusion Tensor Imaging , and correlate these differences with Clinical disability and cognitive disorder results.

DETAILED DESCRIPTION:
The goal of this study is to show pattern differences of vasoreactivity and connectivity between Progressive Multiple Sclerosis and Relapsing Remitting Multiple Sclerosis, by the use of methods of advanced brain MRIs, and correlate these differences with Clinical disability and cognitive disorder results. The modification of the Diffusion Tensor Imaging are well known in these two groups, as well as their link with the occurrence of movement and cognitive disorder. The study of the vasoreactivity during MRI aims to confront our results to the available data sources.

ELIGIBILITY:
Inclusion Criteria :

* For Both patients and healthy volunteers :
* Age limits ≥ 30 et ≤ 50 years
* Subject able to understand the nature, the aim and the methodology of the study.
* Collection of the informed consent
* Affiliation or recipient with the mode of social security.
* For the patients :
* Suffering from progressive multiple sclerosis (primary progressive forms or secondary progressive forms) OR
* Suffering from relapsing-remitting multiple sclerosis

Exclusion Criteria :

* For Both patients and healthy volunteers :
* Systemic pathology with neurological manifestations
* Antecedent of psychiatric disorders including psychosis (Except anxious depressive disorder)
* Subject presenting contraindications in MRI (Ferromagnetic foreign bodies, pace-maker)
* Claustrophobia
* Women pregnant or Breast-feeding
* Person with majority age protected by the law (supervision, trusteeship or under safeguard of justice).
* Subject unable to understand the nature and the aim of the study and/or communication difficulties with investigator
* Antecedent of serious cranial trauma (according to classification) of ischaemic stroke ou intracranial hematoma.
* For the patients :
* Antecedent of serious cranial trauma (according to classification), anterior or evolutive neurologic disease other than multiple sclerosis
* Recent relapse of multiple sclerosis
* For the healthy volunteers :
* Antecedent of serious cranial trauma (according to classification), anterior or evolutive neurologic disease
* Antecedent of neurological disease
* In period of exclusion relative to another protocol or which the annual amount of the allowances maximum of 4500 € was reached.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2017-02-13 (Actual); Study Completion 2017-02-13 (Actual)

PRIMARY OUTCOMES:
Cerebral vasoreactivity measured by diffusion imaging MRI (quantitative variable) :parameter which allow us to estimate the organization of the white matter tracts | 2 months

SECONDARY OUTCOMES:
Comparison of fonctional connective cards at Resting state | 2 months
  somatomotor network and default mode network
Cognitive disorders | 2 months
  Neuropsychological test results (quantitative and quantitative variable)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre LABAUGE, Professor, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Hopital Gui de Chauliac -Service de Neurologie, Montpellier, France